CLINICAL TRIAL: NCT04263324
Title: Beneficial Effects of Self-hypnosis/Self-care Learning Program for Chronic Pain Patients : a MRI and EEG Study
Brief Title: Beneficial Effects of Self-hypnosis/Self-care for Chronic Pain Patients : a MRI and EEG Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Collaborators: Fondation Benoit (Unknown)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Principal Investigator, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/291
Record Dates: First submitted 2020-01-02; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; fibromyalgia; hypnosis; fMRI; EEG
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Each patients will have a medical and a psychological consultation and will have to fill-in questionnaires (T0). Then, they will receive a psycho-education training (5 sessions) and will have to complete the same questionnaires (T1). After that, they will again have a medical (pain doctor) and a psychological consultation. Afterwards, the care staff will have a multidisciplinary discussion about their diagnosis. Then functional Magnetic Resonance Imaging (fMRI; 1 hour) and HdEEG (1 hour) data will be acquired in resting state. After that, participants will receive a 7 months (2 hours session a month) learning program of self-hypnosis/self-care animated by a therapist specialized in hypnosis. After the 7 months learning-program they will complete the same questionnaires (T2) and be scanned again by means of fMRI and HdEEG. Patient who do not want to participate to the learning program will not have a treatment but will be scanned in the fMRI and the HdEEG.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-hypnosis/self-care group (Experimental): It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Self-hypnosis/self-care — Learning phase of self-hypnosis/self-care.
  Arms: Self-hypnosis/self-care group

SUMMARY:
Chronic pain concerns one in four adults in Belgium. Fibromyalgia is an example of chronic pain and is characterized by diffused and migrant musculo-tendinous pain localized in the limbs and at an axial level. The technological improvement in neuroimaging allowed to improve, at a cerebral level, the identification of the structural and the functional characteristics of this clinical entity. Studies indicated a modification in cerebral morphometry showing an alteration of white and grey matter in the anterior cingulate cortex, orbitofrontal lateral cortex, cerebellum, basal ganglia, insula, secondary somatosensory cortex, thalamus, amygdala, putamen, superior temporal gyrus and periaqueductal grey matter. At a functional level, studies show un alteration in the connectivity of the default mode network, an atrophy of zones implicated in nociception and an increased activation of zone implicated in response to a nociceptive stimulus.

Nowadays, researchers are interested in finding out the beneficial effects of non-pharmacological techniques to improve de well-being of patients with chronic pain. Hypnosis is one of these techniques that has already proven to be successful in decreasing pain and improving global quality of life. Nevertheless, to our knowledge, no study has been conducted to understand the impact of hypnosis upon the cerebral functioning of these patients. Therefore, the aim of this study is to understand the impact of a 6 months self-hypnosis/self-care learning program upon the structural and functional functioning of the brain by means of functional magnetic resonance imagery (fMRI) and electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

* Major
* Fluency in French
* Fibromyalgia diagnosis

Exclusion Criteria:

* Neurologic disorder
* Psychiatric disorder
* Drug addiction
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain description | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on pain description will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (no pain) to 10 (worst pain).
Change in sleep difficulties | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care upon the severity of insomnia will be assessed by means of the "Insomnia Severity Index" (Morin et al., 2001). Scale ranging from 0 (none) to 4 (very severe).
Change in anxiety | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on anxiety will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Change in depression | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on depression will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Change in pain disability | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on pain disability will be assessed by means of the "Pain Disability Index" (PDI, Tait et al., 1990). Scale ranging from 0 (no difficulties) to 10 (a lot of difficulties).
Change in attitudes and beliefs about pain | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on the attitudes and beliefs about pain will be assessed my means of the "Survey of Pain Attitudes" (SOPA, Jensen & Karoly, 1987). Scale ranging from 0 (totally wrong) to 10 (totally right).
Change in quality of life | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on the quality of life will be assessed by means of the "Short Form-36"(SF-36; Ware et al., 1988). Each item is balanced to obtain a score between 0 (worst quality) to 100 (maximum quality).
Change in locus of control | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on the locus of control will be assessed my means og the "Multidimensional Health Locus of Control" (MHLC, Wallston et al., 1978). Scale ranging from 1 (no agreement) to 4 (agreement).
Change of the impact of pain | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on the impact of pain in individual's life, quality of social support and general activity, will be assessed my means of the "Multidimensional Pain Index" (PDI, Kerns et al., 1985). Scale ranging from 0 (none) to 6 (a lot).
Change in generic health | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on generic health will be assessed by the "EuroQol 5 Dimensions" questionnaire (EQ-5D, Health Policy, 1990). Scale ranging from 1 (no problems) to 3 (extreme problems).
Change in health status | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of Self-hypnosis/self-care on global health status will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (worst health status) to 100 (best health status).
Change in physical activity | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on the physical activity will be assessed by means of the International Physical Activity Questionnaire (Craig et al., 2003). Participants have to describe the amount of low to intense physical activity they did over a period of 7 days.
Motivation to change | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  The impact of self-hypnosis/self-care on the motivation to change will be assessed by means of the "University of Rhode Island Change Assessment" (URICA, DiClemente et al., 1990). Scale ranging from 1 (no agreement) to 5 (agreement).
Impact on return-to-work | Day 0 (first meeting with the doctor), up to 5 months (before the intervention), up to 12 months (after the intervention)
  For participants who continued to work at time of inclusion, the "Work Design Questionnaire" (WDQ, Morgeson & Hymphrey, 2006) will be administered. Scale ranging from 0 (not at all) to 5 (exactly).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Liège, Liège, Belgium

REFERENCES:
- [Derived] Kumar Govindaiah P, Adarsh A, Panda R, Gosseries O, Malaise N, Salamun I, Tshibanda L, Laureys S, Bonhomme V, Faymonville ME, Vanhaudenhuyse A, Bicego A. Exploring Electrophysiological Responses to Hypnosis in Patients with Fibromyalgia. Brain Sci. 2024 Oct 23;14(11):1047. doi: 10.3390/brainsci14111047. PMID 39595811